CLINICAL TRIAL: NCT06245941
Title: A Phase Ib/II Clinical Trial of TQ05105 Tablets Combined With TQB3909 Tablets in the Treatment of Moderate- and High-risk Myelofibrosis
Brief Title: A Clinical Trial of TQ05105 Tablets Combined With TQB3909 Tablets in the Treatment of Myelofibrosis (MF)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per sponsor request. Premature closure was not prompted by any safety or efficacy concerns.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ05105-TQB3909-Ib/II-01
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-07

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB3909 Tablets (Experimental): TQB3909 Tablets, orally administered. 28 days as a treatment cycle.
  Interventions: Drug: TQB3909 tablets
- TQ05105 Tablets combined with TQB3909 Tablets (Experimental): TQ05105 Tablets combined with TQB3909 Tablets, orally administered. 28 days as a treatment cycle.
  Interventions: Drug: TQ05105 tablets; Drug: TQB3909 tablets

INTERVENTIONS:
Drug: TQ05105 tablets — TQ05105 is a Janus kinase 1 (JAK1) and Janus kinase 2 (JAK2) Inhibitor
  Arms: TQ05105 Tablets combined with TQB3909 Tablets
Drug: TQB3909 tablets — TQB3909 is an inhibitor targeting B-cell lymphoma-2 (BCL-2) protein.

SUMMARY:
This is an open, single-arm, multi-center clinical study designed to evaluate the efficacy and safety of TQ05105 tablets combined with TQB3909 tablets in patients with moderate- and high-risk Myelofibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the study and signed informed consent with good compliance;
* Age: 18 or above (when signing the informed consent form); Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 to 2; Life expectancy ≥ 24 weeks;
* Patients diagnosed with Primary myelofibrosis (PMF), post polycythemia vera myelofibrosis (post-PV-MF), or post essential thrombocythemia myelofibrosis (post-ET-MF);
* Those with moderate or high risk myelofibrosis evaluated according to Dynamic International Prognostic Scoring System (DIPSS) prognostic grading criteria, or those with high risk myelofibrosis according to National Comprehensive Cancer Network (NCCN) guidelines prognostic grading criteria;
* Patients with poor efficacy of JAK inhibitors (for monotherapy of TQB3909, phase Ib and phase II cohort 2);
* Patients who had not received JAK inhibitor treatment (for phase Ib and phase II cohort 2)
* Spleen enlargement;
* Peripheral blood primary cells and bone marrow primary cells are ≤10%;
* No growth factor, colony stimulating factor, thrombopoietin or platelet transfusion was received within 2 weeks before the examination, and the blood routine indexes met the requirements within 7 days before the first administration
* The Main organ function is normal;
* Men and women of childbearing age should agree to use contraceptive measures during the study period and within 6 months after the end of the study.

Exclusion Criteria:

* Patients who have previously received allogeneic stem cell transplantation, or received autologous stem cell transplantation within 3 months before the first administration, or recently planned stem cell transplantation;
* Patients who have previously received BCL-2 inhibitor combined with JAK inhibitor therapy;
* Patients who have previously undergone splenectomy, or received splenic radiotherapy within 6 months before the first administration;
* Other malignancies within 3 years prior to first administration or currently present.
* Patients with multiple factors affecting oral or absorption of drugs;
* Major surgical treatment or significant traumatic injury within 4 weeks prior to first administration;
* Presence of congenital bleeding disorder and congenital coagulopathy;
* Patients who had arterial/venous thrombosis events within 6 months before the first administration.
* Have a history of mental drug abuse, or have a mental disorder.
* Active or uncontrolled severe infection;
* Active hepatitis B virus (HBV) infection, or hepatitis C virus (HCV) infection , or active Corona Virus Disease 2019 (COVID-19) infection;
* Patients with grade III or above congestive heart failure, unstable angina pectoris or myocardial infarction, or arrhythmia requiring treatment, or QT interval prolongation within 6 months before the first administration;
* Unsatisfactory blood pressure control despite standard therapy;
* Patients with renal failure requiring hemodialysis or peritoneal dialysis;
* Patients newly diagnosed with pulmonary interstitial fibrosis or drug-related interstitial lung disease within 3 months before the first administration;
* Patients with a history of immunodeficiency disease or organ transplantation;
* Patients with epilepsy requiring treatment;
* Patients with uncontrolled pleural effusion, pericardial effusion or ascites;
* There is a history of attenuated live vaccine inoculation within 4 weeks before the first administration, or attenuated live vaccine inoculation was planned during the study period.
* People with known hypersensitivity to the study drug and excipients;
* Patients diagnosed as active autoimmune diseases within 2 years before the first administration;
* Those who participated in and used other anti-tumor clinical trial drugs within 4 weeks before the first administration
* Any MF treatment drugs, any immunomodulators, or any immunosuppressants were used within 2 weeks prior to the first dose
* According to the judgment of the investigators, some situations seriously endanger the safety of the subjects or affect the subjects to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Maximal tolerance dose (MTD) | Up to 2 years.
  If dose limiting toxicity (DLT) occurs in 2 or more subjects in a given dose group, the dose level in the previous dose group is considered as MTD.
Recommended phase II dose (RP2D) | Up to 2 years
  The RP2D is defined as the lower dose level to MTD based on the safety profile
35% reduction in spleen volume (SVR35) at week 24 | Up to 24 weeks
  The proportion of subjects with a ≥35% reduction in spleen volume from baseline at the end of treatment at week 24

SECONDARY OUTCOMES:
Optimum effective rate | Up to 120 weeks
  The proportion of subjects with at least once spleen volume reduction ≥ 35% from baseline
Onset time of splenic response | Up to 120 weeks
  The time interval from the first administration to the date when the spleen volume was reduced by ≥ 35 % from baseline
Duration of maintenance of at least 35% Reduction in Spleen Volume (DoMSR) | Up to 120 weeks
  The time between the date when the spleen volume reduction ≥ 35% from baseline occurs for the first time and the date when the spleen volume reduction is < 35% from baseline.
Percentage change in spleen volume from baseline | Up to 60 weeks
  Percentage change in spleen volume of subjects from baseline after treatment.
SVR35 at week 60 | Up to 60 weeks
  The proportion of subjects with a ≥35% reduction in spleen volume compared to baseline after treatment at week 60.
Myeloproliferative neoplasm - Symptom Assessment Form - Total Symptom Score (MPN-SAF-TSS) | Up to 60 weeks
  The proportion of subjects whose total symptom score of MPN-SAF TSS decreased by more than 50% from baseline. MPN-SAF-TSS is a tool for evaluating the disease burden of patients with myeloproliferative neoplasms. Each symptom is scored according to the severity, from asymptomatic (0 points) to the most serious (10 points), a total of 10 levels, the sum of 10 symptom scores is MPN-SAF-TSS score. The higher the score, the more severe the symptoms are.
MPN-SAF-TSS decrease | Up to 60 weeks
  The time and duration when the MPN-SAF-TSS decreased by ≥50% compared to baseline for the first time.
Progression-free survival (PFS) | Up to 120 weeks
  The time interval from the first dose to the date of the occurrence of any of the following events, whichever occurs first:(1) Spleen volume increased by ≥25% compared with the screening period ; (2) Death caused by any cause.
Leukemia free survival (LFS) | Up to 120 weeks
  The time interval from the date of the first dose to the date of any of the following events, whichever occurs first: (1) the date of the first bone marrow smear showing the original cell ≥20% ;(2) The first peripheral blood smear showed that the original cells ≥ 20% and the absolute value of the original cells ≥1×10^9/L and lasted for at least 2 weeks; (3) Death caused by any reason.
Overall Survival (OS) | Up to 120 weeks
  The time from the first time the subject received treatment to death due to any cause
Incidence of adverse events (AEs) | Baseline up to 120 weeks
  Incidence rate of all adverse medical events that occur after the subject receives the investigational drug, evaluated according to the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0)
Severity of adverse events (AEs) | Baseline up to 120 weeks
  Severity of all adverse medical events that occur after the subject receives the investigational drug, evaluated according to the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0)

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - Hennan Cancer Hospital, Zhengzhou, Henan
  - Xijing Hospital of the Fourth Military Medical University, Xi'an, Shaanxi
  - People's Hospital of Tianjin, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital Zhejiang University School Of Medicine, Hangzhou, Zhejiang